CLINICAL TRIAL: NCT00659568
Title: A Phase I Study of Temsirolimus in Combination With Metformin in Advanced Solid Tumours
Brief Title: Metformin and Temsirolimus in Treating Patients With Metastatic or Unresectable Solid Tumor or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CAN-LRCC-UWOREB13877; CDR0000593360 (Registry Identifier: PDQ (Physician Data Query)); WYETH-CAN-LRCC-UWOREB13877
Record Dates: First submitted 2008-04-15; First posted 2008-04-16 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2010-08

CONDITIONS: Breast Cancer; Endometrial Cancer; Kidney Cancer; Lung Cancer; Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent small cell lung cancer; extensive stage small cell lung cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; Waldenström macroglobulinemia
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Kidney Neoplasms; Lung Neoplasms; Lymphoma; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia | interventions — Metformin; temsirolimus

INTERVENTIONS:
Drug: metformin hydrochloride
Drug: temsirolimus

SUMMARY:
RATIONALE: Metformin and temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of metformin when given together with temsirolimus in treating patients with metastatic or unresectable solid tumor or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum tolerated dose and recommended phase II dose of metformin hydrochloride when administered with temsirolimus in patients with advanced solid cancers or lymphoma.

Secondary

* To determine the toxicity and safety, with particular reference to glucose and lipid deregulation, of this regimen in these patients.
* To assess antitumor activity, including tumor response rate and time to progression, in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of metformin hydrochloride.

Patients receive oral metformin once, twice, or three times daily on days 1-28 and temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, including any of the following types:

  * Renal cell
  * Endometrial
  * Breast
  * Small cell lung carcinoma
  * Lymphoma
* Metastatic or unresectable disease for which standard curative or palliative measures do not exist or are no longer effective
* Measurable disease according to RECIST criteria
* No unstable primary CNS tumors or metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* AST ≤ 2.5 times upper limit of normal (ULN)
* Serum creatinine ≤ ULN
* Serum bilirubin ≤ 1.5 times ULN
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to understand and willing to sign a written informed consent document

Exclusion criteria:

* Allergies to or a history of allergic reactions attributed to any other compound of similar chemical or biologic composition to temsirolimus or metformin
* Diabetes mellitus (type I or II)
* Uncontrolled hypertriglyceridemia (triglyceride levels > 10 mmol/L)
* History of lactic acidosis
* Inability to swallow or digest oral medications
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Uncontrolled hypertension
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* Significant traumatic injury within 21 days prior to treatment

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Recovered from all prior therapy
* At least 4 weeks since prior chemotherapy or radiotherapy (6 weeks for carmustine or mitomycin C) except low-dose, non-myelosuppressive radiotherapy
* No limitation on other prior therapy
* Concurrent low-dose anticoagulant (i.e., warfarin) allowed provided INR ≤ 1.1 times ULN
* Concurrent full-dose anticoagulant (i.e., warfarin) allowed provided INR is within institutional therapeutic range (usually 2.0-3.0)

Exclusion criteria:

* Major surgery within the past 21 days
* Prior temsirolimus (or other known inhibitors of mammalian target of rapamycin) or metformin
* Concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent enzyme-inducing anti-epileptic drugs (EIAEDs) (e.g., phenytoin, carbamazepine, or phenobarbital) or other CYP3A4 inducer (e.g., rifampin or Hypericum perforatum [St. John's wort])
* Concurrent investigational or commercial agents or therapies to treat the patient's malignancy
* Other concurrent investigational agents other than temsirolimus or metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-08

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of metformin hydrochloride when administered with temsirolimus

SECONDARY OUTCOMES:
Toxicity and safety, with particular reference to glucose and lipid deregulation
Antitumor activity, including tumor response rate and time to progression
Objective response
Survival
Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mackenzie, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Regional Cancer Program at London Health Sciences Centre, London, Ontario, Canada